CLINICAL TRIAL: NCT01555034
Title: The Effect of Movement Therapy on the Success in a Multidisciplinary Intervention for the Treatment of Childhood Obesity
Brief Title: Movement Therapy and Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 016111CTIL
Record Dates: First submitted 2012-03-08; First posted 2012-03-15 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Obesity
Keywords: obesity; movement therapy; exercise; behaviour
MeSH Terms: conditions — Obesity; Motor Activity; Behavior | interventions — Exercise; Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention plus therapy (Active Comparator)
  Interventions: Behavioral: movement therapy
- intervention no therapy (Active Comparator): exercise and nutrition
  Interventions: Other: exercise plus nutrition

INTERVENTIONS:
Behavioral: movement therapy — exercise, nutrition, movement therapy
  Arms: intervention plus therapy
Other: exercise plus nutrition — exercise, nutrition
  Arms: intervention no therapy

SUMMARY:
The Child health and Sports Center, Meir Medical Center, has an intervention program to treat obese children. The program includes physical activity, nutritional intervention and behavioral treatment.The emphasis given in the center to physical activity and sport enables a strong connection with movement therapy. Movement therapy allows obese children to face and cope with the psychological and emotional aspects of obesity.

The purpose of this study is to evaluate the contribution of the movement therapy intervention to our program.

DETAILED DESCRIPTION:
Movement therapy is part of the multidisciplinary intervention. Weekly one hour long sessions are conducted under the guidance of a certified therapists.

The meeting includes physical movement aimed to address the emotional world of the obese child. Using games, structured exercises and verbal processing.

At the start and end of the evaluation the children will answer questionnaires to study:

1. Behavioral questionnaires:emotional state: anxiety, depression, communication, self-esteem, quality of life and self-efficacy.
2. Demographic questions . At the beginning and the end of the program a certified movement therapist will observe the children to estimate the change of emotional movement.weight, height and BMI are measured regularly in the center.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese children

Exclusion Criteria:

* Child that do not want to take part in this study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2012-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Emotional/behavioral changes | 3 MONTHS
  Change from Baseline in emotional and behavioral questioners at 3 months. The questioners: depression, anxiety, self-efficacy, self-esteem, attachment and quality of life.

SECONDARY OUTCOMES:
weight, height and BMI | 3 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nemet, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel